CLINICAL TRIAL: NCT01787526
Title: High Dose Intravenous Iron in Blood Donors With Iron Deficiency: a Randomized, Controlled Trial
Brief Title: Intravenous High Dose Iron in Blood Donors
Acronym: IronWoMan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0; 2013-000327-14 (EudraCT Number)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Iron Deficiency
Keywords: iron depletion; donor safety; blood donation; transfusion medicine; iron deficiency; intravenous iron; fatigue; restless legs syndrome; anemia
MeSH Terms: conditions — Iron Deficiencies; Fatigue; Restless Legs Syndrome; Anemia | interventions — ferric carboxymaltose; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Iron (Active Comparator): oral iron in a corresponding dose of 10g (assuming an absorption of 10%, 100 capsules a 100mg iron each) taken over 8-12 weeks
  Interventions: Drug: oral iron
- Intravenous high dose iron (Experimental): high dose intravenous iron (ferric carboxymaltose, 1000mg)
  Interventions: Drug: ferric carboxymaltose

INTERVENTIONS:
Drug: ferric carboxymaltose — 1 g intravenously per infusion
  Other Names: ferinject
  Arms: Intravenous high dose iron
Drug: oral iron — oral tablets of 100mg iron over 8 weeks, total dose 10g
  Other Names: Ferretab
  Arms: Oral Iron

SUMMARY:
2-3% of the population participates in blood donation programmes. Traditionally, safety issues in transfusion medicine have been concentrating on product and recipient safety. Extensive efforts including strict donor inclusion criteria and testing for important transmissible infections have substantially improved product quality. One of the most common risks of blood donation is iatrogenic iron deficiency. It may affect up to 30% of regular blood donors because each whole blood donation causes a loss of 200 to 250 mg of iron. Although this has been known for at least 50 years, iron deficiency is not routinely assessed or treated in this population. Contributing factors include donation frequency, lower weight and female gender. Women have lower iron reserves and in premenopausal women, the daily required amount of iron is higher than in men. Besides anemia, iron deficiency may lead to fatigue and impaired cognitive and physical performance. Oral iron substitution is often associated with significant gastrointestinal side effects leading to poor compliance. Today, intravenous (iv.) iron preparations are well tolerated and allow the application of a large dose of 1000mg in one visit. Our hypothesis is that in blood donors with iron deficiency intravenous iron is feasible and preferable to oral iron because of its high efficacy and optimal compliance with a similar safety profile that has been extensively studied in other populations than blood donors.

DETAILED DESCRIPTION:
Iron deficiency is possibly the most prevalent worldwide nutritive deficiency and it has been estimated that > 500 million people have adverse effects as a result. Total body iron amounts to 3 to 4.5 grams, the largest part being bound to hemoglobin in red cells.

One of the most common risks of blood donation is iatrogenic iron deficiency which may affect up to 30% of regular blood donors. Each whole blood donation means a whole blood loss of 450 ml ±10% for the bag and additional samples for the required tests, corresponding to a loss of 200 to 300 mg of iron. It has been estimated that 10 apheresis donations equal 1 whole blood donation. Contributing factors include donation frequency, low body weight and female gender. In Austria, the maximal annual donation frequency is 50x for plasmapheresis, 26x for plateletpheresis and 4 (women) respectively 6x (men) for whole blood donations. Although the frequent donation-induced development of iron depletion has been recognized for at least 50 years, iron deficiency is not routinely assessed or treated in this population. Recently it was reported that the presence of pica, the bizarre consumption of nonnutritive substances such as ice cubes, is associated with a high probability of iron depletion in blood donors.

Contributing factors to a poor iron status in blood donors include donation frequency, lower weight and female gender. Women also have lower iron reserves and in premenopausal women, the daily required amount of iron is higher than in men. Besides anemia, iron deficiency may lead to fatigue and impaired cognitive and physical performance. Several trials have evaluated different regimens of iron substitution in blood donors and demonstrated good treatment compliance and efficacy in improving iron status. Oral iron substitution is often associated with significant gastrointestinal side effects leading to poor compliance. Today, high-dose intravenous (iv.) iron preparations are available, well tolerated and allow for the application of a large dose of 1000mg in one visit.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years and ≤ 65 years
* ferritin ≤ 30 ng/ml
* fulfilment of the strict criteria for blood donation

Exclusion Criteria:

* hemochromatosis
* active infection
* pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
transferrin saturation (%) at visit 1 (V1) | 8 weeks

SECONDARY OUTCOMES:
Number of patients with adverse events of different grades | 8 weeks

OTHER OUTCOMES:
Other parameters of iron metabolism and red blood count | 8 weeks
Subjective symptoms fatigue | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karin Amrein, MD, Principal Investigator — Medical University Graz, Austria
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Background] Amrein K, Valentin A, Lanzer G, Drexler C. Adverse events and safety issues in blood donation--a comprehensive review. Blood Rev. 2012 Jan;26(1):33-42. doi: 10.1016/j.blre.2011.09.003. Epub 2011 Oct 11. PMID 21996651
- [Background] Semmelrock MJ, Raggam RB, Amrein K, Avian A, Schallmoser K, Lanzer G, Semmelrock HJ, Prueller F, Berghold A, Rohde E. Reticulocyte hemoglobin content allows early and reliable detection of functional iron deficiency in blood donors. Clin Chim Acta. 2012 Apr 11;413(7-8):678-82. doi: 10.1016/j.cca.2011.12.006. Epub 2011 Dec 23. PMID 22212625
- [Background] Newman B. Iron depletion by whole-blood donation harms menstruating females: the current whole-blood-collection paradigm needs to be changed. Transfusion. 2006 Oct;46(10):1667-81. doi: 10.1111/j.1537-2995.2006.00969.x. No abstract available. PMID 17002622
- [Background] Cable RG, Glynn SA, Kiss JE, Mast AE, Steele WR, Murphy EL, Wright DJ, Sacher RA, Gottschall JL, Tobler LH, Simon TL; NHLBI Retrovirus Epidemiology Donor Study-II (REDS-II). Iron deficiency in blood donors: the REDS-II Donor Iron Status Evaluation (RISE) study. Transfusion. 2012 Apr;52(4):702-11. doi: 10.1111/j.1537-2995.2011.03401.x. Epub 2011 Oct 24. PMID 22023513
- [Background] Brittenham GM. Iron deficiency in whole blood donors. Transfusion. 2011 Mar;51(3):458-61. doi: 10.1111/j.1537-2995.2011.03062.x. No abstract available. PMID 21388389
- [Background] Bianco C, Brittenham G, Gilcher RO, Gordeuk VR, Kushner JP, Sayers M, Chambers L, Counts RB, Aylesworth C, Nemo G, Alving B. Maintaining iron balance in women blood donors of childbearing age: summary of a workshop. Transfusion. 2002 Jun;42(6):798-805. doi: 10.1046/j.1537-2995.2002.00103.x. No abstract available. PMID 12147035
- [Background] BAST G, PEISKER H, SCHUMANN HD. [Latent disorders caused by iron deficiency in frequent blood donors]. Langenbecks Arch Klin Chir Ver Dtsch Z Chir. 1956;283(3):280-90. No abstract available. German. PMID 13386295
- [Background] Moore RA, Gaskell H, Rose P, Allan J. Meta-analysis of efficacy and safety of intravenous ferric carboxymaltose (Ferinject) from clinical trial reports and published trial data. BMC Blood Disord. 2011 Sep 24;11:4. doi: 10.1186/1471-2326-11-4. PMID 21942989
- [Background] Birgegard G, Schneider K, Ulfberg J. High incidence of iron depletion and restless leg syndrome (RLS) in regular blood donors: intravenous iron sucrose substitution more effective than oral iron. Vox Sang. 2010 Nov;99(4):354-61. doi: 10.1111/j.1423-0410.2010.01368.x. PMID 20598107
- [Derived] Macher S, Herster C, Holter M, Moritz M, Matzhold EM, Stojakovic T, Pieber TR, Schlenke P, Drexler C, Amrein K. The Effect of Parenteral or Oral Iron Supplementation on Fatigue, Sleep, Quality of Life and Restless Legs Syndrome in Iron-Deficient Blood Donors: A Secondary Analysis of the IronWoMan RCT. Nutrients. 2020 May 5;12(5):1313. doi: 10.3390/nu12051313. PMID 32380660
- [Derived] Drexler C, Macher S, Lindenau I, Holter M, Moritz M, Stojakovic T, Pieber TR, Schlenke P, Amrein K. High-dose intravenous versus oral iron in blood donors with iron deficiency: The IronWoMan randomized, controlled clinical trial. Clin Nutr. 2020 Mar;39(3):737-745. doi: 10.1016/j.clnu.2019.03.025. Epub 2019 Mar 26. PMID 30981629
- [Derived] Macher S, Drexler C, Lindenau I, Sareban N, Schlenke P, Amrein K. High-dose intravenously administered iron versus orally administered iron in blood donors with iron deficiency: study protocol for a randomised, controlled trial. Trials. 2016 Oct 28;17(1):527. doi: 10.1186/s13063-016-1648-y. PMID 27793204